CLINICAL TRIAL: NCT02808676
Title: SYNchronizing Exercises, Remedies in GaIt and Cognition (SYNERGIC): A Randomized Controlled Double Blind Trial
Brief Title: SYNchronizing Exercises, Remedies in GaIt and Cognition
Acronym: SYNERGIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the COVID-19 pandemic, in-person interventions/assessments no longer possible.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 107670
Record Dates: First submitted 2016-06-06; First posted 2016-06-22 (Estimated); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognitive training; Vitamin D; Exercise
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Cholecalciferol; Exercise; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Exercises+CognitiveTraining+Vitamin D3 (Experimental): Exercises will combine aerobic+resistance training. Cognitive training will be performed before exercise intervention and using using an "ad-hoc" software developed by us for tablets. Vitamin D3 (10000IU) will be provided orally three time per week for 20 weeks.
  Interventions: Dietary Supplement: Vitamin D3; Other: Exercises (E); Other: Cognitive Training (CT)
- Exercises+CognitiveTraining+Placebo D3 (Experimental): Exercises will combine aerobic+resistance training. Cognitive training will be performed before exercise intervention and using using an "ad-hoc" software developed by us for tablets. Matching placebo of vitamin D3 will be provided orally three time per week for 20 weeks.
  Interventions: Other: Exercises (E); Other: Cognitive Training (CT); Other: placebo D3
- Exercises+Control CogTraining+Vitamin D3 (Experimental): Exercises will combine aerobic+resistance training. Control cognitive training will be performed before exercise intervention and will consist in computer skills training courses. Each session will consist of introductory exercises for computers and different software (e.g., Word, Excel), as well as an initiation to the Internet (search engines, websites, games, etc.). Vitamin D3 (10000IU) will be provided orally three time per week for 20 weeks
  Interventions: Dietary Supplement: Vitamin D3; Other: Exercises (E); Other: control cognitive training
- Exercises+Control CogTraining+Placebo D3 (Experimental): Exercises will combine aerobic+resistance training.Control cognitive training will be performed before exercise intervention and will consist in computer skills training courses. Each session will consist of introductory exercises for computers and different software (e.g., Word, Excel), as well as an initiation to the Internet (search engines, websites, games, etc. Matching placebo of vitamin D3 will be provided orally three time per week for 20 weeks.
  Interventions: Other: Exercises (E); Other: placebo D3; Other: control cognitive training
- Placebo exercise+Control Cog+Placebo D3 (Placebo Comparator): This will be the comparator arm with control/placebo activities.
  Interventions: Other: placebo D3; Other: control cognitive training; Other: Placebo exercise

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Dose: 10000 IU, three times per week, orally.
  Other Names: Cholecalciferol
  Arms: Exercises+CognitiveTraining+Vitamin D3; Exercises+Control CogTraining+Vitamin D3
Other: Exercises (E) — All participants will complete three (3) group training sessions per week (total 20 weeks), under the supervision of trainers. Each exercise session will last approximately 60 minutes and will happen after the cognitive training/control (CT cCT) session. The exercise session will be a combined aerobic and progressive strengthening exercise. Within each small group of four to eight individuals, participants follow the program tailored to their individual functioning level, with constant monitoring by the trainers. Participants are expected to attend all training sessions and research staff will strongly encourage them to do so.
  Arms: Exercises+CognitiveTraining+Placebo D3; Exercises+CognitiveTraining+Vitamin D3; Exercises+Control CogTraining+Placebo D3; Exercises+Control CogTraining+Vitamin D3
Other: Cognitive Training (CT) — CT intervention will involve computer-based multimodal and multi-domain dual-task training with memory load. A custom-written program, developed for neuro-rehabilitation and used in previous research trials for cognitive and mobility outcomes will be used. Training sessions will take place in groups of four to eight participants before each of the fitness-training session for duration of 30 min max. Participants will perform a concurrent visuo-motor task (dual-task combination) composed of different sets of visual stimuli that have to be identified by tapping designated figures on an digital tablet (IOS or Android system). Participants will perform discrimination tasks involving sets of items (e.g. letters, numbers, animals, vehicles, fruits, celestial bodies).
  Arms: Exercises+CognitiveTraining+Placebo D3; Exercises+CognitiveTraining+Vitamin D3
Other: placebo D3 — matching placebo for Vitamin D3
  Arms: Exercises+CognitiveTraining+Placebo D3; Exercises+Control CogTraining+Placebo D3; Placebo exercise+Control Cog+Placebo D3
Other: control cognitive training — As a control activity to ensure the same time exposure as in the interventions arms, participant in the control arm will receive a 30 min computer skills training.
  Arms: Exercises+Control CogTraining+Placebo D3; Exercises+Control CogTraining+Vitamin D3; Placebo exercise+Control Cog+Placebo D3
Other: Placebo exercise — As a control activity to ensure the same time exposure as in the interventions arms, participant in the control arm will receive a 60 min of a tone exercise regimen
  Arms: Placebo exercise+Control Cog+Placebo D3

SUMMARY:
The proposed SYNERGIC trial is uniquely designed to evaluate the effect of aerobic and progressive resistance training exercises, combined with cognitive training and Vitamin D3 supplementation, in cognition and mobility in older adults with Mild Cognitive Impairment (MCI).

DETAILED DESCRIPTION:
Exercises, specifically resistance and aerobic training, have been demonstrated to improve cognitive outcomes, along with improved physical capacity and mobility. Both aerobic and resistance training trials of different duration have revealed positive results, with the most consistent findings being observed after combined interventions of 6 months to one year. Although the training benefits of progressive resistance training (PRT) have been well documented, PRT has been studied far less extensively in older adults with Mild Cognitive Impairment (MCI). Exercise training has proven to be beneficial for cognition even in vulnarable populations like in frail older adults, and those with mobility issues. The exact mechanism supporting the benefits of exercise for cognition in humans needs to be further explored, as numerous studies in animals and humans have demonstrated that aerobic exercise may have neuroprotective and neurorestorative effects. The rationale of combining aerobic and PRT as multimodal exercise intervention is supported by research that has revealed potential beneficial effects. In addition, multimodal exercise interventions have shown positive effects on muscle/lean mass, cognition and brain structure, functionality, and brain volume.

Similarly cognitive training, i.e. computer based cognitive process training, has also shown positive results in improving cognition, mobility, and postural control. Several recent systematic reviews on the topic support the benefits of cognitive training. In line with exercise training, recent research on cognitive training has also supported important improvements in brain plasticity post-intervention.

Finally, Vitamin D3 deficiency in older adults has been linked to cognitive dysfunction, dementia, and mobility decline. Besides its very well-known effects on muscle and bone physiology, several studies have shown a potential beneficial role of Vitamin D3 on cognitive function. Robustly designed trials, with longitudinal follow-up, have been recommended in older adults with MCI to investigate the comparative benefits of isolated Vitamin D3 supplementation, and combined with physical and cognitive training.

To date, the effect of adding cognitive training and/or Vitamin D3 to a multimodal progressive exercise training for improving global cognition, executive function, memory, and gait in MCI has not been assessed.

ELIGIBILITY:
Inclusion Criteria:

1. At least 60 years of age
2. Self-reported levels of proficiency in English (French for Montreal site only) for speaking and understanding spoken language.
3. Able to comply with scheduled visits, treatment plan, and other trial procedures
4. Able to ambulate at least 10 meters independently
5. Having MCI operationalized using Albert et al. criteria as:

   * objective cognitive impairment in one of the following four cognitive domains: memory, executive function, attention, and language evaluated by the Montreal Cognitive Assessment (MoCA) test with scores ranging from 13-24/30.
   * Preserved activities of daily living on the disability scale confirmed by clinician interview
6. Having normal or corrected to normal vision in at least one eye so that they can identify symbols and stimuli presented on a computer screen in front of them.
7. Must be in sufficient health to participate in the study's aerobic-based exercise training program, based on medical history, vital signs, physical examination by study physicians, or written recommendation by family physician indicating one's appropriateness to participate in aerobic-based exercise training program.

Exclusion Criteria:

1. Serious underlying disease (such as active cancer, or recent heart attack) which, in the opinion of the investigator, may preclude engagement in interventions or may interfere with the participant's ability to participate fully in the study.
2. Diagnosis of dementia using criteria from the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition.
3. Participant with uncontrolled major depression, schizophrenia, severe anxiety and substance abuse.
4. Current parkinsonism or any neurological disorder with residual motor deficits (e.g. stroke with motor deficit), active musculo-skeletal disorders (e.g. severe osteoarthritis of lower limbs) or history of knee/hip replacement affecting gait performance at clinical evaluation.
5. Intention to enroll in other clinical trials during the same time period
6. Pre-existing exercise structured training program involving aerobic or resistance training in previous 6 months.
7. Taking cognitive enhancers, neuroleptics, anticholinergics or Vitamin D3 in doses more than 1000IU/day or equivalent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel M Montero-Odasso, MD, PhD, Study Chair — Gait and Brain Lab, Lawson Health Research Institute
Locations (6):
- Canada (6):
  - University of British Columbia, Vancouver, British Columbia
  - St. Joseph's Health Care London, Parkwood Hospital, London, Ontario
  - University of Waterloo, Waterloo, Ontario
  - Wilfrid Laurier University, Waterloo, Ontario
  - Concordia University, Montreal, Quebec
  - Institut Universitaire de Gériatrie de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bherer L, Erickson KI, Liu-Ambrose T. Physical exercise and brain functions in older adults. J Aging Res. 2013;2013:197326. doi: 10.1155/2013/197326. Epub 2013 Sep 17. No abstract available. PMID 24163767
- [Background] Liu-Ambrose T, Nagamatsu LS, Voss MW, Khan KM, Handy TC. Resistance training and functional plasticity of the aging brain: a 12-month randomized controlled trial. Neurobiol Aging. 2012 Aug;33(8):1690-8. doi: 10.1016/j.neurobiolaging.2011.05.010. Epub 2011 Jul 7. PMID 21741129
- [Background] Colcombe S, Kramer AF. Fitness effects on the cognitive function of older adults: a meta-analytic study. Psychol Sci. 2003 Mar;14(2):125-30. doi: 10.1111/1467-9280.t01-1-01430. PMID 12661673
- [Background] Langlois F, Vu TT, Chasse K, Dupuis G, Kergoat MJ, Bherer L. Benefits of physical exercise training on cognition and quality of life in frail older adults. J Gerontol B Psychol Sci Soc Sci. 2013 May;68(3):400-4. doi: 10.1093/geronb/gbs069. Epub 2012 Aug 28. PMID 22929394
- [Background] Sage MD, Almeida QJ. A positive influence of vision on motor symptoms during sensory attention focused exercise for Parkinson's disease. Mov Disord. 2010 Jan 15;25(1):64-9. doi: 10.1002/mds.22886. PMID 19938164
- [Background] Sage MD, Almeida QJ. Symptom and gait changes after sensory attention focused exercise vs aerobic training in Parkinson's disease. Mov Disord. 2009 Jun 15;24(8):1132-8. doi: 10.1002/mds.22469. PMID 19373930
- [Background] Cotman CW, Berchtold NC, Christie LA. Exercise builds brain health: key roles of growth factor cascades and inflammation. Trends Neurosci. 2007 Sep;30(9):464-72. doi: 10.1016/j.tins.2007.06.011. Epub 2007 Aug 31. PMID 17765329
- [Background] Nagamatsu LS, Handy TC, Hsu CL, Voss M, Liu-Ambrose T. Resistance training promotes cognitive and functional brain plasticity in seniors with probable mild cognitive impairment. Arch Intern Med. 2012 Apr 23;172(8):666-8. doi: 10.1001/archinternmed.2012.379. No abstract available. PMID 22529236
- [Background] Kueider AM, Parisi JM, Gross AL, Rebok GW. Computerized cognitive training with older adults: a systematic review. PLoS One. 2012;7(7):e40588. doi: 10.1371/journal.pone.0040588. Epub 2012 Jul 11. PMID 22792378
- [Background] Reijnders J, van Heugten C, van Boxtel M. Cognitive interventions in healthy older adults and people with mild cognitive impairment: a systematic review. Ageing Res Rev. 2013 Jan;12(1):263-75. doi: 10.1016/j.arr.2012.07.003. Epub 2012 Jul 25. PMID 22841936
- [Background] Ballesteros S, Prieto A, Mayas J, Toril P, Pita C, Ponce de Leon L, Reales JM, Waterworth J. Brain training with non-action video games enhances aspects of cognition in older adults: a randomized controlled trial. Front Aging Neurosci. 2014 Oct 14;6:277. doi: 10.3389/fnagi.2014.00277. eCollection 2014. PMID 25352805
- [Background] Chapman SB, Aslan S, Spence JS, Hart JJ Jr, Bartz EK, Didehbani N, Keebler MW, Gardner CM, Strain JF, DeFina LF, Lu H. Neural mechanisms of brain plasticity with complex cognitive training in healthy seniors. Cereb Cortex. 2015 Feb;25(2):396-405. doi: 10.1093/cercor/bht234. Epub 2013 Aug 28. PMID 23985135
- [Background] Annweiler C, Montero-Odasso M, Muir SW, Beauchet O. Vitamin D and Brain Imaging in the Elderly: Should we Expect Some Lesions Specifically Related to Hypovitaminosis D? Open Neuroimag J. 2012;6:16-8. doi: 10.2174/1874440001206010016. Epub 2012 Feb 28. PMID 22423308
- [Background] Beauchet O, Annweiler C, Verghese J, Fantino B, Herrmann FR, Allali G. Biology of gait control: vitamin D involvement. Neurology. 2011 May 10;76(19):1617-22. doi: 10.1212/WNL.0b013e318219fb08. Epub 2011 Apr 6. PMID 21471466
- [Background] Annweiler C, Schott AM, Rolland Y, Blain H, Herrmann FR, Beauchet O. Dietary intake of vitamin D and cognition in older women: a large population-based study. Neurology. 2010 Nov 16;75(20):1810-6. doi: 10.1212/WNL.0b013e3181fd6352. PMID 21079183
- [Background] Montero-Odasso M, Bherer L, Studenski S, Gopaul K, Oteng-Amoako A, Woolmore-Goodwin S, Stoole P, Wells J, Doherty T, Zecevic AA, Galinsky D, Rylett RJ, Jutai J, Muir-Hunter S, Speechley M, Camicioli R. Mobility and Cognition in Seniors. Report from the 2008 Institute of Aging (CIHR) Mobility and Cognition Workshop. Can Geriatr J. 2015 Sep 30;18(3):159-67. doi: 10.5770/cgj.18.188. eCollection 2015 Sep. PMID 26495050
- [Background] Annweiler C, Beauchet O, Bartha R, Hachinski V, Montero-Odasso M; WALK Team (Working group Angers-London for Knowledge). Vitamin D and caudal primary motor cortex: a magnetic resonance spectroscopy study. PLoS One. 2014 Jan 31;9(1):e87314. doi: 10.1371/journal.pone.0087314. eCollection 2014. PMID 24498072
- [Background] Montero-Odasso M, Hachinski V. Preludes to brain failure: executive dysfunction and gait disturbances. Neurol Sci. 2014 Apr;35(4):601-4. doi: 10.1007/s10072-013-1613-4. Epub 2013 Dec 24. PMID 24366243
- [Background] Montero-Odasso M, Verghese J, Beauchet O, Hausdorff JM. Gait and cognition: a complementary approach to understanding brain function and the risk of falling. J Am Geriatr Soc. 2012 Nov;60(11):2127-36. doi: 10.1111/j.1532-5415.2012.04209.x. Epub 2012 Oct 30. PMID 23110433
- [Background] Skinner J, Carvalho JO, Potter GG, Thames A, Zelinski E, Crane PK, Gibbons LE; Alzheimer's Disease Neuroimaging Initiative. The Alzheimer's Disease Assessment Scale-Cognitive-Plus (ADAS-Cog-Plus): an expansion of the ADAS-Cog to improve responsiveness in MCI. Brain Imaging Behav. 2012 Dec;6(4):489-501. doi: 10.1007/s11682-012-9166-3. PMID 22614326
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Fraser SA, Li KZ, DeMont RG, Penhune VB. Effects of balance status and age on muscle activation while walking under divided attention. J Gerontol B Psychol Sci Soc Sci. 2007 May;62(3):P171-8. doi: 10.1093/geronb/62.3.p171. PMID 17507585
- [Background] Montero-Odasso M, Zou G, Speechley M, Almeida QJ, Liu-Ambrose T, Middleton LE, Camicioli R, Bray NW, Li KZH, Fraser S, Pieruccini-Faria F, Berryman N, Lussier M, Shoemaker JK, Son S, Bherer L; Canadian Gait and Cognition Network. Effects of Exercise Alone or Combined With Cognitive Training and Vitamin D Supplementation to Improve Cognition in Adults With Mild Cognitive Impairment: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2324465. doi: 10.1001/jamanetworkopen.2023.24465. PMID 37471089
- [Background] Bray NW, Pieruccini-Faria F, Witt ST, Rockwood K, Bartha R, Doherty TJ, Nagamatsu LS, Almeida QJ, Liu-Ambrose T, Middleton LE, Bherer L, Montero-Odasso M. Frailty and functional brain connectivity (FBC) in older adults with mild cognitive impairment (MCI): baseline results from the SYNERGIC Trial. Geroscience. 2023 Apr;45(2):1033-1048. doi: 10.1007/s11357-022-00702-4. Epub 2022 Dec 21. PMID 36539590
- [Background] Bray NW, Pieruccini-Faria F, Witt ST, Bartha R, Doherty TJ, Nagamatsu LS, Almeida QJ, Liu-Ambrose T, Middleton LE, Bherer L, Montero-Odasso M. Combining exercise with cognitive training and vitamin D3 to improve functional brain connectivity (FBC) in older adults with mild cognitive impairment (MCI). Results from the SYNERGIC trial. Geroscience. 2023 Jun;45(3):1967-1985. doi: 10.1007/s11357-023-00805-6. Epub 2023 May 10. PMID 37162700
- [Derived] Montero-Odasso M, Almeida QJ, Burhan AM, Camicioli R, Doyon J, Fraser S, Li K, Liu-Ambrose T, Middleton L, Muir-Hunter S, McIlroy W, Morais JA, Pieruccini-Faria F, Shoemaker K, Speechley M, Vasudev A, Zou GY, Berryman N, Lussier M, Vanderhaeghe L, Bherer L. SYNERGIC TRIAL (SYNchronizing Exercises, Remedies in Gait and Cognition) a multi-Centre randomized controlled double blind trial to improve gait and cognition in mild cognitive impairment. BMC Geriatr. 2018 Apr 16;18(1):93. doi: 10.1186/s12877-018-0782-7. PMID 29661156

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercises+CognitiveTraining+Vitamin D3: Exercises will combine aerobic+resistance training. Cognitive training will be performed before exercise intervention and using using an "ad-hoc" software developed by us for tablets. Vitamin D3 (10000IU) will be provided orally three time per week for 20 weeks.
  Vitamin D3: Dose: 10000 IU, three times per week, orally.
  Exercises (E): All participants will complete three (3) group training sessions per week (total 20 weeks), under the supervision of trainers. Each exercise session will last approximately 60 minutes and will happen after the cognitive training/control (CT cCT) session. The exercise session will be a combined aerobic and progressive strengthening exercise.
  Cognitive Training (CT): CT intervention will involve computer-based multimodal and multi-domain dual-task training with memory load. A custom-written program, developed for neuro-rehabilitation and used in previous research trials for cognitive and mobility outcomes will be used. Training sessions will take place in groups of four to eight participants before each of the fitness-training session for duration of 30 min max. Participants will perform a concurrent visuo-motor task (dual-task combination) composed of different sets of visual stimuli that have to be identified by tapping designated figures on an digital tablet (IOS or Android system). Participants will perform discrimination tasks involving sets of items (e.g. letters, numbers, animals, vehicles, fruits, celestial bodies).
- Exercises+CognitiveTraining+Placebo D3: Exercises will combine aerobic+resistance training. Cognitive training will be performed before exercise intervention and using using an "ad-hoc" software developed by us for tablets. Matching placebo of vitamin D3 will be provided orally three time per week for 20 weeks.
  Exercises (E): All participants will complete three (3) group training sessions per week (total 20 weeks), under the supervision of trainers. Each exercise session will last approximately 60 minutes and will happen after the cognitive training/control (CT cCT) session. The exercise session will be a combined aerobic and progressive strengthening exercise.
  Cognitive Training (CT): CT intervention will involve computer-based multimodal and multi-domain dual-task training with memory load. A custom-written program, developed for neuro-rehabilitation and used in previous research trials for cognitive and mobility outcomes will be used. Training sessions will take place in groups of four to eight participants before each of the fitness-training session for duration of 30 min max. Participants will perform a concurrent visuo-motor task (dual-task combination) composed of different sets of visual stimuli that have to be identified by tapping designated figures on an digital tablet (IOS or Android system). Participants will perform discrimination tasks involving sets of items (e.g. letters, numbers, animals, vehicles, fruits, celestial bodies).
  placebo D3: matching placebo for Vitamin D3
Period: Overall Study
Arm/Group | Exercises+CognitiveTraining+Vitamin D3 | Exercises+CognitiveTraining+Placebo D3 | Exercises+Control CogTraining+Vitamin D3 | Exercises+Control CogTraining+Placebo D3 | Placebo Exercise+Control Cog+Placebo D3
Started | 34 | 35 | 37 | 35 | 34
Completed | 31 | 28 | 31 | 28 | 26
Not Completed | 3 | 7 | 6 | 7 | 8

BASELINE CHARACTERISTICS:
Population: Participants must be at least 60 years of age, ambulate independently for at least 10 meters, and have a diagnosis of Mild Cognitive Impairment (MCI) based on Albert et al. criteria, including objective cognitive impairment in memory, executive function, attention, or language, MoCA scores between 13-24/30, and preserved activities of daily living confirmed by clinician assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercises+CognitiveTraining+Vitamin D3 | Exercises+CognitiveTraining+Placebo D3 | Exercises+Control CogTraining+Vitamin D3 | Exercises+Control CogTraining+Placebo D3 | Placebo Exercise+Control Cog+Placebo D3 | Total
Number analyzed (Participants) | 34 | 35 | 37 | 35 | 34 | 175
Age, Customized [Count of Participants; unit: Participants] — Population: A total of 175 participants were initially randomized in the study, and baseline characteristics were obtained for all enrolled participants. However, 31 participants withdrew from the study before completing either the intervention or required follow-up assessments and thus were excluded from the final statistical analysis. Data from 144 participants were thus included in the primary statistical analysis.
  Participants
    Age between 65 and 84 years: number analyzed (Participants) | 31 | 28 | 31 | 28 | 26 | 144
    Age between 65 and 84 years | 31 | 28 | 31 | 28 | 26 | 144
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 20 | 12 | 17 | 86
  Male | 13 | 19 | 17 | 23 | 17 | 89
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 34 | 35 | 37 | 35 | 34 | 175

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Cognition Assessed Using the ADASCog(13 and Plus Modalities).
Description: Global cognition will be assessed using the cognitive section of the Alzheimer Disease Assessment Scale-plus EF+FA (ADAS-Cog-plus). This scale consists of 10 brief cognitive tests assessing memory, language, executive function, praxis, and instrumental activities of daily living. The ADAS-Cog has been a significant outcome measure in numerous trials with MCI and AD. The ADAS-Cog-plus has marked advantages as an outcome measure in MCI populations since incorporates items concerning executive function (EF) and functional abilities (FA). Scores in the ADASCog-plus (EF+FA) range from 0 to 90, with higher scores indicating better cognitive performance.
Time Frame: baseline and at 20 weeks (after interventions finalised)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Exercises+CognitiveTraining+Vitamin D3 | Exercises+CognitiveTraining+Placebo D3 | Exercises+Control CogTraining+Vitamin D3 | Exercises+Control CogTraining+Placebo D3 | Placebo Exercise+Control Cog+Placebo D3
Number analyzed (Participants) | 31 | 28 | 31 | 28 | 26
score on a scale | -2.42 (0.70) | -2.14 (0.73) | -0.39 (0.69) | -1.34 (0.73) | 0.24 (0.76)

2. Secondary Outcome: Change in Cognition Assessed as the CCNA Cognitive Battery.
Description: The Canadian Consortium on Neurodegeneration in Aging (CCNA) has established a battery of neuropsychological test which will used as secondary outcomes e.g., ADAS-Cog-13, which is scored from 0 to 70, with higher scores indicating greater cognitive impairment.
Time Frame: baseline at 20 weeks (after interventions finalised)
Measure: Mean (Standard Error); unit: score on a scale (ADAS-Cog-13)
Arm/Group | Exercises+CognitiveTraining+Vitamin D3 | Exercises+CognitiveTraining+Placebo D3 | Exercises+Control CogTraining+Vitamin D3 | Exercises+Control CogTraining+Placebo D3 | Placebo Exercise+Control Cog+Placebo D3
Number analyzed (Participants) | 34 | 35 | 37 | 35 | 34
score on a scale (ADAS-Cog-13) | 15.3 (8) | 14.5 (6.1) | 16.6 (7.6) | 15.6 (6.6) | 13.7 (5.3)

3. Secondary Outcome: Falls Incidence
Description: Frequency and circumstances of falls over the study period.
Time Frame: baseline at 20 weeks (after interventions finalised)
Reporting Status: Not Posted

4. Secondary Outcome: Gait Velocity - cm/s
Description: Assessment of usual and fast-paced walking to evaluate mobility performance.
Time Frame: baseline at 20 weeks (after interventions finalised)
Reporting Status: Not Posted

5. Secondary Outcome: Gait Variability Which is Calculated as Coefficient of Variation (CoV)
Description: A higher CoV indicates greater variability, which has been associated with increased fall risk and impaired motor control, particularly in individuals with Mild Cognitive Impairment (MCI
Time Frame: baseline at 20 weeks (after interventions finalised)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From baseline visit and up to 30 days after study participation has ended month 12 visit.
Arm/Group | Exercises+CognitiveTraining+Vitamin D3 | Exercises+CognitiveTraining+Placebo D3 | Exercises+Control CogTraining+Vitamin D3 | Exercises+Control CogTraining+Placebo D3 | Placebo Exercise+Control Cog+Placebo D3
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35 | 0/37 | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/35 | 1/37 | 2/35 | 0/34
Other Adverse Events (participants affected / at risk) | 8/34 | 12/35 | 9/37 | 13/35 | 6/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercises+CognitiveTraining+Vitamin D3 (N=34) | Exercises+CognitiveTraining+Placebo D3 (N=35) | Exercises+Control CogTraining+Vitamin D3 (N=37) | Exercises+Control CogTraining+Placebo D3 (N=35) | Placebo Exercise+Control Cog+Placebo D3 (N=34)
Minor Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercises+CognitiveTraining+Vitamin D3 (N=34) | Exercises+CognitiveTraining+Placebo D3 (N=35) | Exercises+Control CogTraining+Vitamin D3 (N=37) | Exercises+Control CogTraining+Placebo D3 (N=35) | Placebo Exercise+Control Cog+Placebo D3 (N=34)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 4 (4) | 8 (8) | 3 (3)
Fall (tripped or slipped) (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Numbness (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dizziness (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Others (General disorders) | 1 (1) | 4 (4) | 3 (3) | 2 (2) | 1 (1) — Systolic blood pressure readings too high, knee pain, hip pain, back pain, chest discomfort, pressure in the head, profuse sweating, headache, head injury in garage, pneumonia, shingles, herpes zoster.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT02808676/Prot_SAP_000.pdf